CLINICAL TRIAL: NCT05999578
Title: Evaluating the Contribution of Hypnosis on Image Quality During Cardiac Magnetic Resonance Imaging (MRI) in Anxious Patients
Brief Title: Contribution of Hypnosis on Image Quality in Cardiac MRI
Acronym: HYPNOLINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2022/79
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Anxiety
Keywords: hypnosis; cardiac MRI; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anxious patients with hypnosis (Experimental): Hypnosis support before, during and at the end of cardiac MRI exam
  Interventions: Other: Hypnosis
- Anxious patients without hypnosis (No Intervention): Cardiac MRI exam accordingly to usual care
- Non anxious patients (No Intervention): Cardiac MRI exam accordingly to usual care

INTERVENTIONS:
Other: Hypnosis — Hypnosis support before, during and at the end of cardiac MRI exam
  Arms: Anxious patients with hypnosis

SUMMARY:
The present project aims to explore the effect of a hypnosis session performed on a patient with anxiety during a cardiac MRI examination on image quality.

DETAILED DESCRIPTION:
Cardiac Magnetic Resonance Imaging (MRI) is an activity of the Bordeaux University Hospital that continues to grow (+7.3% in 2021 compared to 2019) under the combined effect of the increase in activity of cardiology care channels and the extension of clinical indications for cardiac MRI. Indeed, cardiac MRI has become an essential examination in the diagnosis of many heart diseases and is little practiced elsewhere in New Aquitaine. The current delay for a cardiac MRI is 3 and a half months.

In this context, it is necessary to be efficient because any procedure failure, examination interruption or insufficient image quality can delay the diagnosis and therapeutic management of the patient for several months. Numerous studies have shown that anxiety induces interruptions in the acquisition of MRI images and repetition of sequences, thus prolonging the examination time.

However, no study takes into account the specificity of cardiac MRI, whose image quality is intimately linked to the patient's cooperation and to the synchronization of the sequences with the heart rhythm.

Hypnosis seems to be adapted to reduce the patient's anxiety, by allowing him to ignore the surrounding reality while remaining in relation with the attendant.

The hypothesis is that by reducing patient anxiety through hypnosis, image quality in cardiac MRI would be improved.

ELIGIBILITY:
Inclusion Criteria:

* Anxious patient (anxiety score TRAIT (baseline) and anxiety score STATE (situational) ≥ 46) and non-anxious patient (anxiety score TRAIT and anxiety score STATE < 46) requiring cardiac MRI for diagnosis or follow-up of a cardiac pathology except the patients with cardiac arrhythmias or irregular heartbeats.
* 18 years and older
* Highly effective contraception for women of childbearing potential, maintained during research procedures
* Informed consent
* Affiliated or beneficiary of health insurance

Exclusion Criteria:

* Contraindications to MRI and gadoline contrast medium
* Hearing impaired patients
* Patients who do not speak French
* Women who are pregnant or lactating
* Inability to agree to participate to the study
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
quality of cardiac MRI images | Baseline
  Likert score measurements

SECONDARY OUTCOMES:
number of artifacts | Baseline
  The number of artifacts will be estimated with European CMR Registry objective score.
Diagnostic validation score | Baseline
  The diagnostic validation score for the entire examination (and not sequence by sequence) makes it possible to define whether, despite the presence of artifacts, the examination makes it possible to answer the question initially asked in the examination request.
Causality score measurement | Baseline
  Causality score measurement for examinations with a Likert score < 4
Overall duration | Baseline
  The overall duration of the examination and the different phases (reception and preparation time, image acquisition time).
Number of repeated or interrupted sequences | Baseline
  The number of repeated or interrupted sequences (by the Radiographer or the patient).
Anxiety level | Baseline
  The Spielberg State Anxiety Index STAI-Y anxiety score will be used to estimate patient anxiety before and after the MRI.
Post-MRI satisfaction score | Baseline
  The post-MRI satisfaction score will be estimated from the patient by a visual analog scale rated from 0 (not at all satisfied) to 10 (very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No